CLINICAL TRIAL: NCT06194565
Title: Molecular Imaging of HER2 Expression in Breast Cancer Using 99mTc-ABH2 SPECT/CT
Brief Title: 99mTc-ABH2 SPECT/CT in Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-ABH2
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 99mTc-ABH2 SPECT/CT (Experimental): The patients will be injected with 5.55 to 7.4 MBq per kilogram body weight of 99mTc-ABH2 in one dose intravenously and undergo SPECT/CT scan 1h to 2h later.
  Interventions: Drug: 99mTc-ABH2

INTERVENTIONS:
Drug: 99mTc-ABH2 — Each patient will receive an intravenous injection of 99mTc-ABH2, and undergo a SPECT/CT scan within specified time.

SUMMARY:
This prospective study will investigate the potential usefulness of 99mTc-ABH2 SPECT/CT in the diagnostic performance and evaluation efficacy of breast cancer.

DETAILED DESCRIPTION:
This study aims to assess the diagnostic performance of 99mTc-ABH2 SPECT/CT for the detection of HER2-positive primary breast cancer and possible metastases. Visual and semiquantitative methods will be utilized to evaluate the acquired SPECT/CT images. A comparative analysis of tumor imaging data and HER2 expression obtained by immunohistochemistry (IHC) and/or fluorescent in situ hybridization (FISH) analysis of biopsy samples will further be conducted. Results of HER2 expression imaging may have potential significance in screening and monitoring individuals for targeted therapy with monoclonal antibodies, like Trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* clinically suspected primary breast cancer by mammography or ultrasonography and being able to sign the written informed consent form

Exclusion Criteria:

* pregnancy or lactation, impaired liver or kidney failure, and undergoing any preceding local or systemic therapies that might interfere HER2 binding

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
SPECT/CT-based 99mTc-ABH2 uptake value in tumor lesions | 1 year
  Uptake of 99mTc-ABH2 in the lesions will be assessed using SPECT/CT and measured in standardized uptake value (SUV).

CONTACTS AND LOCATIONS:
Overall Officials: Hongli MD Jing, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China